CLINICAL TRIAL: NCT05982262
Title: Naturopathic-pharmacological Consultation on the Use of Dietary Supplements in Patients With Hematological Diseases
Brief Title: Naturopathic-pharmacological Consultation in Hematology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0149-20-BNZ
Record Dates: First submitted 2023-07-16; First posted 2023-08-08 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Hematologic Diseases
Keywords: Dietary supplements; Herbal supplements; Hematology; Safety; Consultation; Naturopath; Clinical pharmacist
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with hematological conditions (Experimental): Patients will be referred by the medical or nursing staff of the Hematology Unit at the Bnai Zion Medical Center according to inclusion criteria
  Interventions: Other: Naturopathic-pharmacological consultation

INTERVENTIONS:
Other: Naturopathic-pharmacological consultation — The naturopathic-pharmacological consultation includes a naturopath and a clinical pharmacist and will consist of at least two meetings.

SUMMARY:
The goal of this cross-sectional study is to learn about the effect of a naturopathic-pharmacologic consultation in patients with hematologic conditions. The main question it aims to answer is whether such consultation can improve the safety of dietary and herbal supplements' use among these patients.

Participants will be asked to answer basic questions and fill-out questionnaire before and after meeting the consultation team. Some patients will be prescribed dietary and herbal supplements that may help relief some of the symptoms they describe, in a safe way and without interacting with the drugs they are taking.

ELIGIBILITY:
Inclusion Criteria:

1. Followed up for a hematological condition
2. Ability to fill simple questionnaires in Hebrew, Russian or Arabic
3. Indication for consultation:

   1. Patient's request to expand knowledge about the use of DHS
   2. Patient using DHS
   3. Patient's desire to start using DHS
   4. Patient that is interested in hearing about the use of DHS for his/her health condition
   5. Medical or nursing team's recommendation to take DHS for medical treatment or to improve compliance with conventional treatment.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Safety of the use of DHS in patients with a hematological disease through naturopathic counseling | From enrollment to the end of intervention, up to 1 year
  Number of potential interactions with moderate to major level of significance prevented by the naturopathic consultation in each patient, as well as the incidence of DHS-related safety events. The Naranjo and modified Food and Drug Administration algorithm will be used to assess the causality of such events with the specific dietary supplements, and only side effects at least possibly caused by the DHS according to these scales will be considered.

SECONDARY OUTCOMES:
Efficacy of prescribed dietary and herbal supplements (DHS) | From enrollment to the end of intervention, up to 1 year
  Measure Yourself Concerns and Wellbeing (MYCAW) questionnaire: requires participants to nominate one or two concerns and, using a seven-point scale from 0 (worse outcome) to 6 (best outcome), to score these concerns and their general feeling of wellbeing.
Patient-physician communication around the use of DHS | From enrollment to the end of intervention, up to 1 year
  Asking the patient whether the topic has been brought up with the treating hematologist and checking the documentation of the use of DHS in the medical charts
Patient satisfaction | From enrollment to the end of intervention, up to 1 year
  Direct question asked after each meeting ranking in a 1-5 Likert scale the satisfaction of the patient from the consultation: from 1 (not satisfied at all) to 5 (maximal satisfaction)
Compliance with hematological treatment | From enrollment to the end of intervention, up to 1 year
  Relative dose intensity (RDI) of the prescribed hematological drugs both before and after intervention: The term of dose intensity (DI) is used to define the drug dose delivered per time unit and is expressed as mg/m2 per week. A delay in the sequence of treatment cycles decreases the DI in the same proportion as a reduction of dose. Average relative DI corresponds to the mean DI of combined agents and is expressed as a fraction of a similar combination selected as a standard
Qualitative evaluation of the staff and patients from naturopathic-pharmacological counseling | From enrollment to the end of intervention, up to 1 year
  Semi-structured in-depth interviews will be conducted with patients who are interested in participating in the qualitative arm (10-15 patients) and the staff members involved (medical staff, nursing staff, naturopath, clinical pharmacist). The goal is to describe the process of building the naturopathic-pharmacological consultation and evaluate the satisfaction of the staff and patients

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Levy Yurkovski, MD, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT05982262/Prot_SAP_001.pdf